CLINICAL TRIAL: NCT04859972
Title: Adherence of Primary Care Doctors to Guidelines of Making a Positive Diagnosis of IBS.
Brief Title: How Well do Primary Care Doctors in Region Örebro County, Sweden Follow Diagnostic Guidelines of IBS?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 277069
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Rome IV; Functional gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with IBS: Patients diagnosed with IBS within primary care in Region Örebro County between 2015- 2019, identified by ICD-code K.58.
  Interventions: Diagnostic Test: Diagnosis of IBS

INTERVENTIONS:
Diagnostic Test: Diagnosis of IBS — Diagnosis of IBS according to ICD-10

SUMMARY:
The aim of this project is to investigate the implementation of the Rome criteria in daily primary care clinical practice and adherence of general practitioners (GPs) to recommended diagnostic approaches for IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disorder. To diagnose IBS, the so-called Rome Criteria combined with limited laboratory tests should be used. However, within the primary care, too much unnecessary diagnostics, for example radiology and endoscopy, are used. This is meaningless, stressful for the patient and they also cost a lot of money.

In Örebro Region there are 29 public general health centers. Approximately 300.000 inhabitants are listed within these health centers. Approximately 150 doctors are currently working within the primary health care of Örebro Region. The software program Medrave and the electronic patient register in Örebro Region allows to search for the International Statistical Classification of Diseases (ICD-10) for IBS (K58.9 and K58.0) This allows retrospective research regarding diagnosing IBS, the used diagnostic tools, comorbidities, as well as the different treatments that were used.

Patients diagnosed with IBS will be identified by ICD-code K.58. By evaluating their patient register it will be determined how the GP has made the IBS diagnosis. Patients will fall into three categories: those who received a positive IBS diagnosis using the Rome criteria, those who received a negative IBS diagnosis and those whose patient record is lacking sufficient information.

Data will also include demographics, number of GP contacts and referrals to specialists, diagnostic procedures, treatments, and relevant somatic, psychological and psychiatric comorbidities. Data regarding substance abuse will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

• All adult patients (both sexes) who were diagnosed with IBS according to ICD-10 in Region Örebro County 2015-2019.

Exclusion Criteria:

• Patients < 18 years or > 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IBS within primary care of Region Örebro County 2015-2019.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-22 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to guidelines of making a positive diagnosis of IBS within primary care. | 2015-2019
  The proportion of patients that received a positive IBS diagnosis versus the proportion of patients that received a negative IBS diagnosis.

SECONDARY OUTCOMES:
Prevalence of diarrhea-predominant IBS and IBS without diarrhea. | 2015-2019
  Proportion of patients with diarrhea-predominant IBS versus IBS without diarrhea
The proportion of IBS patients that have one or more comorbidities. | 2015-2019
  Data will be collected about the following comorbidities: depression (F32, F33 and F41.2), anxiety (F41), somatization syndrome (F45), posttraumatic stress syndrome (F43.1), sleeping disorder (G47.9), urinary incontinence (N39.3 and N39.4), fecal incontinence (R15.9), migraine (G43), headache (R51.9 and G44.2), menstruation symptoms (N92 and N94), fibromyalgia (M79.7), Ehlers Danlos syndrome (Q79.6), other unspecific muskuloskeletal pain (M79) and functional dyspepsia (K30.9).
The proportion of IBS patients with post-infectious IBS. | 2015-2019
  The presence of gastroenteritis (A09.9) that precedes the diagnosis of IBS.
The proportion of IBS patients with substance abuse. | 2015-2019
  Data will be collected regarding substance abuse which is defined by alcohol (F10), opioids (F11), cannabis (F12), sedatives and hypnotics (F13) and Tobacco (F17).

CONTACTS AND LOCATIONS:
Overall Officials: Michiel van Nieuwenhoven, Associate Professor, M.D. PhD., Principal Investigator — Region Örebro County